CLINICAL TRIAL: NCT02274090
Title: Local Drug Delivery of 1% Metformin Gel in Moderate and Severe Periodontitis Subjects: a Randomized Controlled Clinical Trial
Brief Title: 1% Metformin in Moderate and Severe Periodontitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Government Dental College and Research Institute, Bangalore (Other)
Responsible Party: Principal Investigator, Dr. A R Pradeep, Professor, Government Dental College and Research Institute, Bangalore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GDCRI/ACM/PG/PhD/10B/2013-14
Record Dates: First submitted 2014-10-17; First posted 2014-10-24 (Estimated); Last update posted 2014-10-24 (Estimated); Status verified 2014-10

CONDITIONS: Periodontitis
Keywords: Metformin; Pocket depth; moderate periodontitis; severe periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo Group (Placebo Comparator): Placebo gel without the active ingredient. Delivered in biodegradable gel. Frequency- One dose each at baseline, 3 month and 6 month.
  Interventions: Drug: Placebo gel
- 1% Metformin (Active Comparator): 1% Metformin gel. Delivered in biodegradable gel. Frequency- One dose each at baseline, 3 month and 6 month.
  Interventions: Drug: 1% Metformin gel

INTERVENTIONS:
Drug: Placebo gel — Placebo gel consist of drug without the active component.
  Other Names: Placebo group
  Arms: Placebo Group
Drug: 1% Metformin gel — Metformin gel consist of active component.
  Other Names: 1% Metformin group
  Arms: 1% Metformin

SUMMARY:
This study evaluates the efficacy of 1% Metformin gel in treatment of moderate and severe periodontitis subject.

DETAILED DESCRIPTION:
Metformin (MF) has stimulating effect of osteoblastic lineages. In the present study seventy subjects were categorized into two treatment groups: Scaling and root planing (SRP) plus 1% MF and SRP plus placebo. Clinical parameters were recorded at baseline, 3, 6 and 9 months; they included plaque index (PI), modified sulcus bleeding index (mSBI), probing depth (PD), and clinical attachment level (CAL). Radiologic assessment of intra bony defect (IBD) and percentage defect depth reduction (DDR%) was done at baseline, 6 months and 9 months interval using computer-aided software. PD, CAL and defect depth reduction was evaluated in initial pocket depth of ≥5mm and ≥7mm subgroup within placebo and MF group.

Mean probing depth reduction and mean clinical attachment level gain was found to greater in MF group than placebo group at all visits. Significantly greater mean percentage of defect depth reduction was found in MF group than the placebo sites in both ≥5mm and ≥7mm of initial periodontal pocket depth. In MF group improvement in clinical parameter were similar in both the sites, with slightly better improvement in clinical parameters in initial pocket depth ≥7mm with respect to CAL, IBD and DDR% while PD was significantly reduced in initial pocket depth of ≥7mm.

There was greater decrease in mSBI and PD and more CAL gain with significant IBD depth reduction at the sites treated with SRP plus locally delivered MF in chronic periodontitis subjects with intrabony defects as compared to placebo and effect of MF was similar in initial moderate periodontal pockets and deep pocket depths.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy subjects, Pocket depth ≥ 5 mm, Clinical attachment level ≥ 4 mm and vertical bone loss ≥ 3 mm on intraoral periapical radiographs, with no history of periodontal therapy in the last 6 months.

Exclusion Criteria:

* subjects allergic to MF, those on systemic MF therapy, subjects with aggressive periodontitis, immunocompromised subjects, use of tobacco in any form, alcoholics, lactating and pregnant females.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2013-11; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Percentage reduction in Defect depth | at 6 months and 9 months

SECONDARY OUTCOMES:
Plaque index | at 3 , 6 and 9 months
Modified sulcular bleeding index | at 3 , 6 and 9 months
Pocket depth | at 3 , 6 and 9 months
Clinical attachment level | at 3 , 6 and 9 months

REFERENCES:
- [Derived] Pradeep AR, Patnaik K, Nagpal K, Karvekar S, Guruprasad CN, Kumaraswamy KM. Efficacy of 1% Metformin Gel in Patients With Moderate and Severe Chronic Periodontitis: A Randomized Controlled Clinical Trial. J Periodontol. 2017 Oct;88(10):1023-1029. doi: 10.1902/jop.2017.150096. Epub 2017 Jul 21. PMID 28731373